CLINICAL TRIAL: NCT05874804
Title: A Clinical Study With the Carry Life® UF System in Continuous Ambulatory Peritoneal Dialysis (CAPD) Patients
Brief Title: Carry Life@ UF System Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Triomed AB (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Tmed-010; CIV-23-03-042555 (Other: Medical Products Agency, Sweden)
Record Dates: First submitted 2023-04-18; First posted 2023-05-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-10

CONDITIONS: End Stage Renal Disease
Keywords: Steady concentration peritoneal dialysis; SCPD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control CAPD treatment (Active Comparator): The subjects will receive their standard CAPD treatment.
  Interventions: Drug: 2.27% glucose peritoneal dialysis dwell
- Carry Life UF (Experimental): Three days per week, the subject will replace a 2.27% glucose dwell with the Carry Life® UF treatment. The remaining four days of the week, one 2.27% glucose dwell will be replaced by a 1.36% glucose dwell.
  Interventions: Device: Carry Life UF

INTERVENTIONS:
Device: Carry Life UF — A 5-hour treatment with the Carry Life UF used with a 1.36% glucose PD fill.
  Arms: Carry Life UF
Drug: 2.27% glucose peritoneal dialysis dwell — A 5-hour CAPD dwell with a 2.27% glucose PD fluid.
  Arms: Control CAPD treatment

SUMMARY:
The Carry Life UF system performs peritoneal ultrafiltration by adding glucose to the low glucose strength (1.36%) peritoneal dialysis fluid which has been instilled into the peritoneal cavity prior to the connection of the device. By maintaining a stable glucose concentration in the intraperitoneal fluid during the 5-hour treatment, the ultrafiltration can be increased compared to a standard CAPD dwell.

DETAILED DESCRIPTION:
A study of the peritoneal ultrafiltration achieved with Carry Life® UF system compared to standard peritoneal dialysis (PD) therapy, in CAPD patients.

The study consists of the following five (5) phases:

1. Inclusion phase.
2. In-clinic treatment phase for dose determination and safety evaluation.
3. Randomization phase.
4. Transition to home treatment phase.
5. Home treatment phase for efficacy and safety evaluation.

The in-clinic phase consists of one 2.27% Peritoneal equilibrium test (PET) and two Carry Life® UF treatments; one with a 11 g/h glucose dose and one with a 15 g/h glucose dose. The Carry Life® UF treatments will be used for a safety evaluation and based on the UF volumes achieved with the Carry Life® UF treatments, the Carry Life® UF glucose dose for the home treatment phase will be determined. A 24-h urine sample will be collected before the first visit for determination of residual renal function.

After completion of the in-clinic treatment phase, subjects will be randomized to start the home treatment phase either with the control treatment arm or with the Carry Life® UF treatment arm. Subjects in the control arm will continue their standard CAPD treatment as prescribed. In the Carry Life® UF arm, for three days of the week one 2.27% glucose CAPD dwell per day will be replaced by a Carry Life® UF treatment. For the remaining four days of the week, one 2.27% glucose CAPD dwell will be replaced with a 1.36% glucose CAPD dwell.

Immediately before the subject starts using the Carry Life® UF device at home, there will be a transition to the home treatment phase during which the subjects will undergo training on the device and an assessment of their device competency will be performed.

During the home treatment phase of the study, the subject will record body weight, blood pressure and heart rate daily in a patient diary. The PD fill and drain volumes for each dwell during the study will be recorded, as well as any clinical symptoms or device malfunctions.

At the start of the second and third week of each study arm of the home treatment phase a nurse will contact the subject to check on clinical status, AEs, and Carry Life® UF device malfunctions.

Based on the clinical assessments throughout the study, the responsible physician will adjust the subject's PD prescription in order to maintain an adequate fluid balance according to clinical judgement and standard clinical practice. In the control arm, the glucose concentration of the PD dwells may be adjusted as required.

Efficacy evaluation days: The efficacy evaluation days will be performed during week 2 and week 4 of each study arm during the home treatment phase.

During the efficacy evaluation days the dialysate drained from the comparator 2.27% glucose dwell (control) and from the Carry Life® UF treatment will be collected by a research assistant for endpoint evaluation. The 2.27% glucose control dwell will be 5 hours i.e., the same duration as the Carry Life® UF treatment.

The day after the completion of each arm (control and Carry Life® UF), the subject will visit the clinic for data collection. A 24-hour urine sample will be collected before each end-of-arm visit for determination of residual renal function.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Subjects with ESKD treated with PD for at least three (3) months.
3. A PD prescription of 2-4 CAPD dwells/day unchanged for a minimum of two (2) weeks, with at least one 1.5-2L, 2.27% glucose day dwell daily.
4. Subjects must be able to tolerate a 2 L PD fill volume for the PET.
5. Subjects using the Baxter PD system with a MiniCap transfer set.
6. In the opinion of the Investigator, the subject has the capacity to learn how to use the Carry Life® UF system or has a caregiver who can do so.
7. Obtained written consent to participate in the study.

Exclusion Criteria:

1. A PD prescription including a regular 3.86% glucose day dwell.
2. An episode of peritonitis within the last three (3) months.
3. Serum potassium > 6 mmol/l within the last three (3) months.
4. Serum urea > 35 mmol/l within the last three (3) months.
5. Clinical signs of dehydration.
6. Systolic blood pressure < 100 mmHg within the last month.
7. Known diagnosis of clinically significant aortic stenosis.
8. Clinical condition of unstable diabetes.
9. Subjects with a life expectancy of < six (6) months.
10. Evidence of any other diseases or medical conditions that may interfere with the planned treatment or affect participant compliance.
11. Participation in clinical trials, interfering with the present study, within the previous month.
12. Anticipated living donor kidney transplantation within six (6) months of screening.
13. Pregnant, breastfeeding, or women of childbearing potential who are not using an effective method of contraception (hormonal contraceptives or barrier contraceptive methods).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Ultrafiltration volume | 8 weeks
  The UF volume is the difference between the drained fluid volume and the administered fluid volume. The average of two treatments per arm during the home phase of the study.

SECONDARY OUTCOMES:
Adverse event rates | 8 weeks
  Rates of adverse events (AEs) and serious adverse events (SAEs) during the home phase of the study.
Peritoneal sodium removal | 8 weeks
  Sodium removed with the drained fluid volume minus the sodium administered with the PD fluid. The average of two treatments per arm during the home phase of the study.
Glucose UF efficiency | 8 weeks
  ml UF/gram glucose absorbed.Glucose absorbed is the glucose added with the solutions minus the glucose removed by the peritoneal drains. The average of two treatments per arm during the home phase of the study
Peak dialysate glucose concentration | 2 weeks
  The peak glucose concentration recorded during the two Carry Life UF treatments in the clinic phase of the study.

OTHER OUTCOMES:
Peritoneal urea and creatinine removal | 8 weeks
  The amount of the urea and creatinine removed by the peritoneal drains. The average of two treatments for each arm during the home phase of the study.
Weekly peritoneal ultrafiltration volume | 8 weeks
  Based on the PD diary. The sum of the UF volumes from all dwells during each study week during the home phase of the study

CONTACTS AND LOCATIONS:
Overall Officials: Olof Heimbürger, MD, PhD, Principal Investigator — Karolinska Institutet; Stanley Fan, MD, PhD, Principal Investigator — Barts & The London NHS Trust; Giuseppe Castellano, MD, PhD, Principal Investigator — Policlinic of Milan, Italy
Locations (11):
- Italy (2):
  - ASST-Cremona, Cremona
  - Polyclinic Milan, Milan
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Skånes University Hospital, Lund
  - Karolinska Universitetssjukhuset, Njurmedicin Rosenlund, Stockholm
- United Kingdom (6):
  - Heartlands Hospital, Birmingham
  - Queen Elisabeth's Hospital, Birmingham
  - King's College Hospital, London
  - London Royal Hospital, Barth Health NHS Trust, London
  - Royal Free London NHS Foundation Trust, London
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilkie M, de Leon C, Carlsson O, Hegbrant J, Heimburger O. A clinical study of efficacy and safety of the Carry Life UF system in continuous ambulatory peritoneal dialysis patients: protocol for a prospective, multicenter, randomized, crossover study. BMC Nephrol. 2025 Apr 3;26(1):174. doi: 10.1186/s12882-025-04095-2. PMID 40181271

DOCUMENTS (1):
  • Study Protocol (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT05874804/Prot_000.pdf